CLINICAL TRIAL: NCT04489225
Title: Personalized Therapy Study - Heart Failure Risk Status (TriageHF) Post Approval Study
Brief Title: Personalized Therapy Study - HFRS (TriageHF) Post Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: HFRS PAS
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: This single arm observational study includes all patients implanted with a Medtronic Cobalt™ XT ICD or CRT-D MRI SureScan™ (with Attain StabilityQuad™ MRI SureScan™ Model 4798 Lead (ASQ)), who are enrolled in the Medtronic CareLink (CL) Network and Product Surveillance Registry (PSR). Patients will be followed per the standard of care practices of their care provider. All patients must provide a signed informed consent.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational only without any intervention

SUMMARY:
Medtronic is sponsoring the HFRS PAS to evaluate the HFRS feature (TriageHF) when used in routine clinical practice following commercial release. The HFRS PAS is conducted within Medtronic's Product Surveillance Registry (PSR) platform.

DETAILED DESCRIPTION:
The HFRS PAS is a global, prospective, observational, multi-site study. Patients implanted with a Medtronic Cobalt™ XT CRT (with Attain StabilityQuad™ MRI SureScan™ Model 4798 Lead (ASQ)) or ICD device who are enrolled in the Medtronic CareLink (CL) Network and the PSR will be followed per the standard of care practices of their care provider.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible ICD or CRT device or Patients may be enrolled pre-implant and up to 30 days post-implant following confirmation of patient eligibility.
* Patient is enrolled in the Medtronic CareLink® Network for remote monitoring.

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes all patients implanted with a Medtronic Cobalt™ XT ICD or CRT-D MRI SureScan™ (with Attain StabilityQuad™ MRI SureScan™ Model 4798 Lead (ASQ)), who are enrolled in the Medtronic CareLink (CL) Network and Product Surveillance Registry (PSR).
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
positive predictive value (PPV) of HFRS High Risk Status associated with worsening heart failure | Up to 5 years
  To estimate the positive predictive value (PPV) of HFRS High Risk Status associated with worsening heart failure

SECONDARY OUTCOMES:
Number of HF hospitalization or HF related deaths | Up to 5 years
  Summarize the number of HF hospitalization or HF related deaths that were not preceded by a High-Risk Status.

CONTACTS AND LOCATIONS:
Locations (92):
- United States (51):
  - Southwest EP, Chandler, Arizona
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Chula Vista Cardiac Center, Chula Vista, California
  - Cardiovascular Consultants Medical Group, Van Nuys, California
  - Cardiology Associates Medical Group, Ventura, California
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - Denver Heart, Denver, Colorado
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Have, Connecticut
  - Heart Rhythm Solutions, Hollywood, Florida
  - Baptist Health, Jacksonville, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Heart Rhythm Consultants P.A. (Sarasota Memorial Research), Sarasota, Florida
  - Deaconess Specialty Physicians, Evansville, Indiana
  - Iowa Heart, Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Norton Heart and Vascular Institute, Louisville, Kentucky
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - Associates in Cardiology PA, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University Hospital of Missouri, Columbia, Missouri
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medicine, Omaha, Nebraska
  - Monmouth Cardiology Associates, Eatontown, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - Huntington Hospital, Huntington, New York
  - North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York-Presbyterian Hospital/Weill-Cornell Medical Center, New York, New York
  - NewYork-Presbyterian/Columbia University Irving Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Staten Island University Hospital, Staten Island, New York
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Summa Center for Clinical Trials-Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Christ Hospital Health Network, Cincinnati, Ohio
  - St Lukes University Health Network, Bethlehem, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Consultants in Cardiology, Fort Worth, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- France (11):
  - Clinique Rhone Durance, Avignon, France
  - Ch de La Region D'Annecy, Metz-Tessy, France
  - Nouvelles Cliniques Nantaises, Nantes, France
  - Chu Nord Saint-Étienne, Saint-Priest-en-Jarez, France
  - CHU de Brest, Brest
  - CHU de Caen - Hôpital Côte de Nacre - Centre Esquirol, Caen
  - Générale de Santé - Hôpital Privé Saint Martin, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - CHU de Dijon - Hospital Le Bocage, Dijon
  - CHRU La Rochelle, La Rochelle
  - Capio - Clinique du Tonkin, Villeurbanne
- Greece (2):
  - Hygeia Hospital, Athens
  - Athens Medical Center, Marousi
- Italy (6):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Sanitaria Provinciale di Cosenza "Ospedale di Castrovillari", Cosenza
  - Ospedale "Vito Fazzi" Lecce, Lecce
  - Azienda Ospedaliera Ospedale Niguarda Ca Granda, Milan
  - Presidio Ospedaliero Centrale - SS. Annunziata, Taranto
  - Azienda ospedaleria Santa Maria della Misericordia di Udine, Udine
- Portugal (4):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Hospital de Santa Maria-Centro Hospitalar Lisboa Norte, EPE, Lisbon
  - Centro Hospitalar Universitário de São João, Porto
  - Hospital Distrital de Santarém, Santarém
- Národný ústav srdcových a cievnych chorôb, a.s. (NÚSCH, a.s.), Bratislava, Slovakia
- Spain (8):
  - Hospital Universitario da Coruña, A Coruña
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Cardiopark Zurich, Zurich
- United Kingdom (7):
  - University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - Blackpool, Fylde and Wyre Hospitals NHS Foundation Trust - Blackpool Victoria Hospital, Blackpool
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - Central Manchester University Hospitals NHS - Manchester Royal Infirmary, Manchester
  - The James Cook University Hospital - South Tees Hospitals NHS, Middlesbrough
  - Sheffield Vascular Institute, Sheffield Teaching Hospitals NHS - Northern General, Sheffield